CLINICAL TRIAL: NCT04735237
Title: Philtrum Reconstruction Using Autogenous Fat Injection Versus a Surgical Repair With Orbicularis Reconstruction, in Secondary Unilateral Cleft Lip Revision (A Randomized Clinical Trial)
Brief Title: Philtrum Reconstruction Using Autogenous Fat Injection Versus a Surgical Repair in Secondary Unilateral Cleft Lip Revision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Shereen Ishak Faris, Assistant Researcher, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Omfs 3.3.8
Record Dates: First submitted 2021-01-19; First posted 2021-02-03 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Unilateral Cleft Lip
Keywords: Cleft lip; Unilateral Cleft lip; Lip revision surgery; Secondary lip repair; Autogenous fat injection
MeSH Terms: conditions — Cleft Lip | interventions — Reoperation

STUDY DESIGN:
Intervention Model Description: * A randomized controlled clinical trial.
  * The trial will be carried out in the clinic of Oral and Maxillofacial Surgery Department- Faculty of Dentistry-Cairo University & Pediatric Plastic Surgery Department (clinic & operative theatre), Cairo University.
  * Equal randomization: participants with equal probabilities for randomization.
  * Parallel group study: Each group of patient receives a single treatment simultaneously.
Who Masked: Participant, Outcomes Assessor
Masking Description: Each patient will be given a code by the main researcher and the raters will be blind to which group this case belongs. Patients, raters and statistician will be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous fat injection (Experimental): Fat will first be harvested from the abdomen, then injected into the lip
  Interventions: Procedure: Autogenous fat injection
- Surgical revision with orbicularis oris muscle reconstruction (Active Comparator)
  Interventions: Procedure: Surgical revision with orbicularis oris muscle reconstruction.

INTERVENTIONS:
Procedure: Autogenous fat injection — Done under general anesthesia. Fat is to be harvested from the abdomen using manual liposuction. Small aliquots of fat are to be injected into the philtral column (and in the vermilion and any other area of volume insufficiency if needed).
  Arms: Autogenous fat injection
Procedure: Surgical revision with orbicularis oris muscle reconstruction. — Surgical repair done under general anesthesia. The original scar will be marked on the skin with methylene blue. The skin will be incised along the designed line with scar removal. The orbicularis oris muscle stump will be dissected medially and laterally and approximated by means of 4-0 inverted horizontal mattress sutures.
  Other Names: Secondary cleft lip revision surgery
  Arms: Surgical revision with orbicularis oris muscle reconstruction

SUMMARY:
Two groups of patients with repaired unilateral cleft lip deformity having mild to moderate grooving and/or scarring of the philtral column and requiring a secondary cleft lip repair.

* The first group will receive upper lip fat injections into the philtral column (and other areas of volume insufficiency if needed) after manual fat liposuction from the abdomen.
* The second group will receive surgical lip revision with reconstruction of the orbicularis oris muscle using inverted horizontal mattress sutures for enhancement of the philtral ridge.

DETAILED DESCRIPTION:
Interventions:

A. Intervention group: Fat injection

Harvesting fat from the donner site:

1. Surgical repair is to be done under general anesthesia.
2. IV infusion of cephalosporine antibiotic as surgical prophylaxis against infection
3. Tumescent fluid of normal saline and epinephrine 1:500,000 is to be hand infiltrated into the donor site (abdomen).
4. The lipoaspirate is to be harvested from the donor site using manual liposuction through a small incision (less than 0.5 cm). Fat is aspirated using a blunt tipped catheter on a 10-mL syringe.
5. The fat is emulsified.

Injecting fat into the lip:

1. The micro fat is reloaded into a 1-mL syringe and injected with a 1.5 mm blunt-tipped grafting needle.
2. Small aliquots of fat are injected into the philtral column.
3. Fat is to be injected in the vermilion and any other area of volume insufficiency if needed, depending on the contour of the lip.

B. Comparator group: Surgical revision with orbicularis oris muscle reconstruction.

1. Surgical repair is to be done under general anesthesia.
2. IV infusion of cephalosporine antibiotic as surgical prophylaxis against infection
3. The original scar will be marked on the skin with methylene blue.
4. The operating area will be injected with 0.5% lidocaine (containing 1:200,000 epinephrine).
5. The skin will be incised along the designed line with scar removal.
6. The orbicularis oris muscle stump is to be dissected medially and laterally.
7. In the medial segment, the dissection is restricted to within 5 mm medially to avoid crossing the center of the philtral dimple and to prevent any disruption of the normal philtral dimple. The muscle on the lateral cleft segment is to be freed from skin and mucosal by scissor dissection.
8. The medial and lateral orbicularis oris muscle stumps are approximated by means of 4-0 inverted horizontal mattress sutures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with repaired unilateral cleft lip deformity.
2. Mild to moderate grooving and/or scarring of the philtral column.
3. Patients who require a secondary cleft lip repair.
4. Age of the patient between 4 & 16 years
5. All patients are free from any systemic disease that may affect normal tissue healing.

Exclusion Criteria:

1. Patients older than 16 years old or whose caregivers declined a revisionary operation.
2. Patients with any systemic disease that may affect normal healing.
3. Patients with any other craniofacial malformation.
4. Syndromic cleft patients.

Ages: 4 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy of fat injection (or lip revision surgery) in philtral column enhancement assessed by measuring change in philtral column height using photographs and scores of a visual analogue sale (VAS). | preoperative, immediate postoperative, after one year.
  Change in philtral column height as assessed using photographs and scores of a visual analogue scale (scale described below).
  1. Same height as the normal side
  2. Less prominent than the normal side
  3. Flat philtral column
  4. Slight groove
  5. Prominent groove ( lesser scores mean better outcomes and higher scores mean worse outcomes)
Efficacy of fat injection (or lip revision surgery) in philtral column enhancement assessed by measuring change in philtral column projection in mm using a special device clinically. | preoperative, immediate postoperative, after one year.
  Change in philtral column projection as assessed clinically using a special device to obtain quantitative measurements of philtral column projection in mm.
Efficacy of fat injection (or lip revision surgery) in philtral column enhancement assessed by measuring change in height and projection of philtral column in mm using lip ultrasonography. | preoperative, immediate postoperative, after one year.
  Change in height and projection of philtral column as assessed using lip ultrasonography to obtain quantitative measurements of philtral column height and projection in mm.

SECONDARY OUTCOMES:
Efficacy of fat injection (or lip revision surgery) in scar tissue modulation measured by assessing change in the appearance of the scar using photographs and scores of a VAS preoperatively, immediately postoperative and after one year. | preoperative, immediate postoperative, after one year
  Change in the appearance of the scar as assessed by photographs and scores of a three point visual analogue scale (scale described below).
  1. Significantly better than preoperative status
  2. No significant changes
  3. Widened scar ( lesser scores mean better outcomes and higher scores mean worse outcomes)
Satisfaction of patient after lip injection (or lip revision surgery) as assessed by scores of a patient's satisfaction survey. | After one year
  Patient's satisfaction survey (range: 0-20 points).

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Abdel-Ghany, PhD, Study Director — Cairo University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogers CR, Meara JG, Mulliken JB. The philtrum in cleft lip: review of anatomy and techniques for construction. J Craniofac Surg. 2014 Jan;25(1):9-13. doi: 10.1097/SCS.0b013e3182a2dce4. PMID 24240763
- [Background] Cho BC, Baik BS. Formation of philtral column using vertical interdigitation of orbicularis oris muscle flaps in secondary cleft lip. Plast Reconstr Surg. 2000 Oct;106(5):980-6. doi: 10.1097/00006534-200010000-00003. PMID 11039367
- [Background] Kim SW, Oh M, Park JL, Oh AK, Park CG. Functional reconstruction of the philtral ridge and dimple in the repaired cleft lip. J Craniofac Surg. 2007 Nov;18(6):1343-8. doi: 10.1097/scs.0b013e31814e07de. PMID 17993879
- [Background] Fan Q, Li Y, Danning Z, Zhang B, Chen S, Wang J. "Three-unit" muscle reconstruction in secondary cleft lip repair. Cleft Palate Craniofac J. 2015 Jan;52(1):88-95. doi: 10.1597/13-048. PMID 24443976
- [Background] Li L, Xie F, Ma T, Zhang Z. Reconstruction of Philtrum Using Partial Splitting and Folding of Orbicularis Oris Muscle in Secondary Unilateral Cleft Lip. Plast Reconstr Surg. 2015 Dec;136(6):1274-1278. doi: 10.1097/PRS.0000000000001795. PMID 26595020
- [Background] Yin N, Song T, Wu J, Chen B, Ma H, Zhao Z, Wang Y, Li H, Wu D. Unilateral microform cleft lip repair: application of muscle tension line group theory. J Craniofac Surg. 2015 Mar;26(2):343-6. doi: 10.1097/SCS.0000000000001460. PMID 25723667
- [Background] Naidoo S, Butow KW. Philtrum reconstruction in unilateral cleft lip repair. Int J Oral Maxillofac Surg. 2019 Jun;48(6):716-719. doi: 10.1016/j.ijom.2018.11.003. Epub 2018 Dec 7. PMID 30501933
- [Background] Wei J, Deng N, Herrler T, Zhang Y, Li Q, Hua C, Dai C. Short term results of philtrum reconstruction with an orbicularis oris muscle flap in cleft patients. J Craniomaxillofac Surg. 2020 Jun;48(6):569-573. doi: 10.1016/j.jcms.2020.03.008. Epub 2020 Apr 7. PMID 32340907
- [Background] Ma H, Zhang N, Yin N, Guo B. Application of a Layered Muscle Flap Technique for the Reconstruction of the Cupid's Bow and Vermilion in the Repair of Secondary Cleft Lip Deformities. J Craniofac Surg. 2019 Nov-Dec;30(8):e723-e727. doi: 10.1097/SCS.0000000000005714. PMID 31261342
- [Background] Lim AA, Allam KA, Taneja R, Kawamoto HK. Constructing the philtral column in the secondary cleft lip deformity: utilizing the palmaris longus graft. Ann Plast Surg. 2013 Mar;70(3):296-300. doi: 10.1097/SAP.0b013e3182326ef3. PMID 23038138
- [Background] Wang Y, Qi Z, Wang X. Dermis reconstruction and dermis fat graft through an intraoral incision: a new method to correct the furrowed philtral column deformity in lesser-form cleft lip. Cleft Palate Craniofac J. 2014 Mar;51(2):184-8. doi: 10.1597/12-076. Epub 2013 Jan 15. PMID 23320841
- [Background] Nadjmi N, Amadori S, Van de Casteele E. Secondary Cleft Lip Reconstruction and the Use of Pedicled, Deepithelialized Scar Tissue. Plast Reconstr Surg Glob Open. 2016 Oct 25;4(10):e1061. doi: 10.1097/GOX.0000000000001061. eCollection 2016 Oct. PMID 27826467
- [Background] Diepenbrock RM, Green JM 3rd. Autologous Fat Transfer for Maxillofacial Reconstruction. Atlas Oral Maxillofac Surg Clin North Am. 2018 Mar;26(1):59-68. doi: 10.1016/j.cxom.2017.11.002. Epub 2017 Dec 8. No abstract available. PMID 29362072
- [Background] Jones CM, Mackay DR. Autologous Fat Grafting in Cleft Lip and Palate. J Craniofac Surg. 2019 May/Jun;30(3):686-691. doi: 10.1097/SCS.0000000000005205. PMID 31048606
- [Background] Zheng D, Zhou J, Yu L, Zhang Y, Wang J. Autologous Fat Transplantation to Improve Lip Contour in Secondary Cleft Lip Deformity. J Craniofac Surg. 2020 Mar/Apr;31(2):343-346. doi: 10.1097/SCS.0000000000006071. PMID 31856127
- [Background] Koonce SL, Grant DG, Cook J, Stelnicki EJ. Autologous Fat Grafting in the Treatment of Cleft Lip Volume Asymmetry. Ann Plast Surg. 2018 Jun;80(6S Suppl 6):S352-S355. doi: 10.1097/SAP.0000000000001348. PMID 29401128
- [Background] Alighieri C, Bettens K, Roche N, Bruneel L, Van Lierde K. Lipofilling in patients with a cleft lip (and palate) - a pilot study assessing functional outcomes and patients' satisfaction with appearance. Int J Pediatr Otorhinolaryngol. 2020 Jan;128:109692. doi: 10.1016/j.ijporl.2019.109692. Epub 2019 Sep 20. PMID 31568953
- [Background] Jones CM, Morrow BT, Albright WB, Long RE, Samson TD, Mackay DR. Structural Fat Grafting to Improve Reconstructive Outcomes in Secondary Cleft Lip Deformity. Cleft Palate Craniofac J. 2017 Jan;54(1):70-74. doi: 10.1597/15-197. Epub 2016 Jan 11. PMID 26752128
- [Background] Chang FC, Wallace CG, Hsiao YC, Huang JJ, Liu CS, Chen ZC, Chen PK, Chen JP, Chen YR. Long-term comparison study of philtral ridge morphology with two different techniques of philtral reconstruction. Int J Oral Maxillofac Surg. 2020 Oct;49(10):1254-1259. doi: 10.1016/j.ijom.2020.01.015. Epub 2020 Jan 30. PMID 32007356
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair: a double-blinded, randomized, vehicle-controlled clinical trial. PLoS One. 2014 Dec 26;9(12):e115690. doi: 10.1371/journal.pone.0115690. eCollection 2014. PMID 25541942
- [Background] Zhang WH, Chen YY, Liu JJ, Liao XH, Du YC, Gao Y. Application of ultrasound imaging of upper lip orbicularis oris muscle. Int J Clin Exp Med. 2015 Mar 15;8(3):3391-400. eCollection 2015. PMID 26064229